CLINICAL TRIAL: NCT05984693
Title: The Effect of Video-Assisted Instruction on the Ability of Midwifery Students to Provide Health Education
Brief Title: Video-Assisted Instruction and Health Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Döndü BATKIN ERTÜRK, Assist. Prof. Dr, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: TOKAT03
Record Dates: First submitted 2023-07-22; First posted 2023-08-09 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Educational Problems
Keywords: Video-Assisted Instruction; Health Education; Skill; Midwifery student
MeSH Terms: conditions — Health Education

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Experimental group students determined by randomization will be shown videos containing examples of health education prepared by the researchers. After watching each video, the right and wrong aspects of health education will be critically evaluated, discussed with the group, and the group's suggestions for improving education will be taken.
  Interventions: Behavioral: Video Assisted Instruction
- Control groups (No Intervention): Control group students will not receive any training other than theoretical training.

INTERVENTIONS:
Behavioral: Video Assisted Instruction — Video Assisted Instruction
  Arms: Experimental group

SUMMARY:
This research was conducted to examine the effect of video-assisted teaching on the health education skill of midwifery students.

DETAILED DESCRIPTION:
Despite emphasizing the importance of the role of health professionals as health educators, it is observed that health professionals assigned with health education mostly behave in line with their personal abilities and experiences while training on health-related issues. However, in order for health education to reach its goals, what health education is, its role in health promotion should be understood correctly, the principles of health education, the planning and implementation steps of health education should be well known. The effectiveness of the nurse as an educator depends on her feeling herself equipped in the role of educator and having gained knowledge, skills, attitudes and behaviors related to education. A nurse's ability to teach effectively can optimize patients' knowledge, skills, self-care abilities, and ability to make informed choices. In a study, it was reported that the knowledge, skills and attitudes of nurses regarding health education competence were low, and the main factors affecting the health education practice were lack of education and training, lack of time and workload. In another study, from the point of view of nursing students, lack of knowledge, lack of communication skills and heavy workload were reported as the main obstacles to patient education. Similarly, another study found that health education and health promotion skills of health professionals are generally not at an acceptable level.Teaching patients effectively requires knowledge and skill. Nurses can develop their teaching/teaching skills through practice, training and mentoring. Therefore, the development of health education skills of midwives, who have important roles and responsibilities in the protection and development of maternal and newborn, women's and community health, is important for them to fully fulfill these roles and responsibilities.

Today, technology has become an indispensable part of the teaching process and has always played an important role in skills training. Video-based learning refers to knowledge or skills acquired through video-based instruction. Video is a tool that appeals to more sense organs because it provides the opportunity to use image and sound together and is used for modeling. The use of videos in educational environments has effects such as cognitive benefit (learning a lot and well, keeping in memory, remembering), psychological benefits (motivation, learning pleasure) and ease of visualizing information. The use of video in the learning process helps students to create meaningful mental activities and to develop cognitive abilities such as interpretation, critical thinking, and problem-solving skills. The literature supports the use of video as a teaching method in gaining psychomotor skills to midwifery and nursing students. According to our current knowledge, no study has been found in the national and international literature on the ability of midwives to provide health education. In this study, the effect of video-assisted instruction on midwifery students' ability to give health education was examined. It is thought that the data obtained from this study will contribute to the literature on this subject and will be a source of inspiration for new studies.

Place and Time: The research was conducted in Tokat Gaziosmanpaşa University, Faculty of Health Sciences, Midwifery Department, between 01/04/2023-01/07/2024.

Population and Sample of the Research: The population of the research consisted of second-year students (n=88) who took the "Teaching in Midwifery" course in the 2022-2023 academic year, spring semester at Tokat Gaziosmanpaşa University, Faculty of Health Sciences, Department of Midwifery.

The sample of the randomized controlled study was calculated in the G*Power 3.1 program. According to this, the number of samples to be included in the study for an 80% statistical power 0.05 margin of error was calculated as n=44 for the experimental group and n=44 for the control group for each group. Students were assigned to the groups by adding them to the first column of the Microsoft Excel program according to the sequence number in the list and deriving the number in the second column. In the study, 1 represents the experimental group and 0 represents the control group.

Characteristics of Participants Data Collection: The subjects of the Midwifery Education course in the spring semester of the 2022-2023 academic year were taught theoretically by the responsible lecturers of the course to the 2nd grade midwifery students included in the research. All the students included in the research were asked to identify any health education topic, to prepare a teaching plan and original educational material for the subject. The research group was asked to fill out the "Question Form on the Effect of Video Assisted Instruction on the Health Education Skills of Midwifery Students". The students in the experimental group determined by randomization were shown the videos containing the health education example prepared by the researchers. After watching each video, the right and wrong aspects of health education will be critically evaluated, discussed with the group, and the group's suggestions for improving education were received. The control group students did not receive any training other than theoretical training. One week later, all students in the research group were asked to present the health education they had prepared for the topic they determined, using materials, to a peer in the classroom environment in about 10 minutes. All students' health education skills were evaluated by the researchers according to the "Health Education Skills List for the Healthy/Sick Individual". When the research data is completed, the applications will be made by the researchers to all students in the control group in order to ensure equality of opportunity in education.

Data Collection Tools

1. "The Effect of Video Assisted Instruction on Health Education Skills of Midwifery Students Questionnaire"
2. "Health Education Skills List for Healthy/Sick Individuals"

In the skill list, each process step was evaluated as "adequate", "development and insufficient", "adequate" was scored as 2, "development" was scored as 1 and "insufficient" was scored as 0.

Analysis of Data Descriptive statistics will be calculated to give information about the general characteristics of the research groups. Qualitative data will be shown as numbers and percentages, Chi-Square Test or Fisher Exact Tests will be used for comparisons between groups. Quantitative data will be shown with mean and standard deviation, Independent Two-Sample T-Test or Mann-Whitney U-Test will be used for comparisons of quantitative data between groups. When p values are calculated below 0.05, they will be considered statistically significant. Calculations will be made with ready-made statistical software. The research will be conducted in accordance with the principles of the Declaration of Helsinki. Permission will be obtained from the institution where the research will be conducted.

Dependent Variables: Students' health education experience and "Health education skill score for the Healthy/Sick Individual"

Independent Variables: Students' socio-demographic characteristics

ELIGIBILITY:
Inclusion Criteria:

All students enrolled in the Teaching in Midwifery (Compulsory) course in the 2nd year curriculum of the Midwifery Department

Exclusion Criteria:

Students who did not volunteer to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Health Education Skills List for Healthy/Sick Individuals | up to 1 month
  In the skill list, each process step was evaluated as "adequate" 2 points, "must be improved" 1 point and "inadequate" 0

CONTACTS AND LOCATIONS:
Overall Officials: Döndü BATKIN ERTÜRK, AssistProfDr, Study Director — Tokat Gaziosmanpasa University
Locations (1):
- Tokat Gaziosmanpasa University, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hacıalioğlu N (2009). Sağlık Eğitimi, Erci B (Edt) Halk Sağlığı Hemşireliği, Göktuğ Yayıncılık, Amasya, Ss: 166-181
- [Background] Hacıalioğlu N (2019). Hemşirelikte Öğretim, Öğrenme ve Eğitim Sağlık Eğitimi, Nobel Tıp Kitapevleri, İstanbul, Ss: 97-108
- [Background] Babacan E, Alıcı S.U. (2008). Hemşirelerin hasta eğitimi ile ilgili düşünce ve uygulamaları. Koç Üniversitesi Hemşirelikte Eğitim ve Araştırma Dergisi (HEAD), 5(2), 29-36.
- [Background] Flanders, S. A. (2018). Effective patient education: Evidence and common sense. Medsurg Nursing, 27(1), 55-58.
- [Background] Pueyo-Garrigues M, Pardavila-Belio MI, Canga-Armayor A, Esandi N, Alfaro-Diaz C, Canga-Armayor N. NURSES' knowledge, skills and personal attributes for providing competent health education practice, and its influencing factors: A cross-sectional study. Nurse Educ Pract. 2022 Jan;58:103277. doi: 10.1016/j.nepr.2021.103277. Epub 2021 Dec 15. PMID 34929565
- [Background] Ghorbani R, Soleimani M, Zeinali MR, Davaji M. Iranian nurses and nursing students' attitudes on barriers and facilitators to patient education: a survey study. Nurse Educ Pract. 2014 Sep;14(5):551-6. doi: 10.1016/j.nepr.2014.06.003. Epub 2014 Jun 26. PMID 25023615
- [Background] Kabasakal, E., & Kublay, G. (2017). Health education and health promotion skills of health care professionals working in family health centres. International Journal of Medical Research & Health Sciences, 6(3).
- [Background] Sablić, M., Mirosavljević, A. & Škugor, A. Video-Based Learning (VBL)-Past, Present and Future: an Overview of the Research Published from 2008 to 2019. Tech Know Learn 26, 1061-1077 (2021). https://doi.org/10.1007/s10758-020-09455-5 Accessed 23 Feb 2023.
- [Background] Korhan, E. A., Tokem, Y., Yılmaz, D. U., Dilemek, H. (2016). Hemşirelikte psikomotor beceri eğitiminde video destekli öğretim ve OSCE uygulaması: bir deneyim paylaşımı. İzmir Kâtip Çelebi Üniversitesi Sağlık Bilimleri Fakültesi Dergisi, 1(1), 35-37.
- [Background] Seferoğlu SS(2013). Öğretim Teknolojileri ve Materyal Tasarımı. 7. Baskı. Pegem Akademi, Ankara, ss:98-102
- [Background] Clerkin R, Patton D, Moore Z, Nugent L, Avsar P, O'Connor T. What is the impact of video as a teaching method on achieving psychomotor skills in nursing? A systematic review and meta-analysis. Nurse Educ Today. 2022 Apr;111:105280. doi: 10.1016/j.nedt.2022.105280. Epub 2022 Jan 24. PMID 35139443
- [Background] Coyne E, Rands H, Frommolt V, Kain V, Plugge M, Mitchell M. Investigation of blended learning video resources to teach health students clinical skills: An integrative review. Nurse Educ Today. 2018 Apr;63:101-107. doi: 10.1016/j.nedt.2018.01.021. Epub 2018 Jan 31. PMID 29425738